CLINICAL TRIAL: NCT01337492
Title: Pilot Study: Safety and Feasibility of Using Sorafenib as Neoadjuvant Treatment Prior to Orthotopic Liver Transplantation (OLT) in Patients With Hepatocellular Carcinoma
Brief Title: Pilot Study Sorafenib as Bridge to Orthotopic Liver Transplantation (OLT)
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: Bayer (Industry); Onyx Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2209
Record Dates: First submitted 2011-01-19; First posted 2011-04-19 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Hepatocellular Carcinoma; Orthotopic Liver Transplant
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental)
  Interventions: Drug: Nexavar

INTERVENTIONS:
Drug: Nexavar — 400 mg of Sorafenib

SUMMARY:
Patients with either histological confirmation or clinical diagnosis who are candidate for orthotopic liver transplant(OLT) will receive Sorafenib 400mg 2 x day (BID) as a neoadjuvant (bridging) treatment until transplant. If patient progresses or falls outside of the Milan criteria on sorafenib patient can be treated per physician's discretion using local therapy. Patient will be followed until 30 days after the orthotopic liver transplant (OLT).

DETAILED DESCRIPTION:
Primary objective:

• To evaluate safety (including possible surgical complication) and feasibility of using sorafenib as neo-adjuvant (bridging therapy) prior to orthotopic liver transplant(OLT).

The primary goal of this pilot study is to assess the safety and feasibility of treating HCC patients with sorafenib prior to OLT, as determined by the number of patients experiencing grade 4 hemorrhaging or bleeding post-operatively.

To achieve these goals a 2-stage accrual design will be used with a maximum accrual goal of 10 patients. Initially 5 patients will be entered on-study. If more than one patient experiences grade 4 hemorrhaging/bleeding following OLT the trial will be closed and sorafenib will not be considered safe and/or feasible. If no patient experiences this event 5 additional patients will be enrolled. At the end of the study sorafenib will be considered safe and feasible in this setting if no patient experience grade 4 hemorrhaging/bleeding following transplant. With this design, and assuming at least 3 of the 5 patients in each cohort undergo OLT, the likelihood of stopping early is <.04 if the underlying risk hemorrhages/bleeding are low (<5% each) whereas there is a >.42 chance of early termination if the risks are substantial (e.g. >.20 likelihood of dose limiting toxicity and >.30 likelihood of >grade 4 hemorrhages/bleeding). Overall the likelihood of accepting or not accepting sorafenib as safe and feasible are >.84, and <.16, respectively under these conditions.

Secondary objectives:

* Drop out rate
* Time to progression prior to orthotopic liver transplant (OLT)
* Waiting time.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years old
* Confirmation of diagnosis of Hepato Cellular Carcinoma (HCC) and within Milan criteria awaiting liver transplant or going through evaluation for Liver Transplant.
* Either histological confirmation or clinical diagnosis by American Association for the Study of Liver Diseases(AASLD) criteria (see Appendix 1) in cirrhotic subjects is required. For subjects without cirrhosis histological confirmation is mandatory.
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Child Pugh A or B (Total point of 7 will be allowed See appendix for scoring system). (ONLY 4 patients with Child Pugh B7 will be allowed.)
* Adequate bone marrow, liver and renal function as assessed by the following:
* Hemoglobin > 8.5 g/dl
* Absolute neutrophil count (ANC) > 1,500/mm3
* Platelet count > 60,000/mm3
* Total bilirubin < 1.5 times Upper Limits of Normal (ULN)
* ALT and AST < 2.5 times the Upper Limits of Normal (ULN) ( < 5 x ULN for patients with liver involvement)
* Creatinine < 1.5 times Upper Limits of Normal (ULN)
* Women of childbearing potential must have 2 negative serum pregnancy test performed. The first test within 7-10 days prior to the start of treatment. The second test within 24 hours prior to start of treatment.
* Women of childbearing potential and men must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation. Men should use adequate birth control for at least three months after the last administration of sorafenib.
* Ability to understand and the willingness to sign a written informed consent. A signed informed consent must be obtained prior to any study specific procedures.

Exclusion Criteria

* Cardiac disease: Congestive heart failure > class II New York Heart Association (NYHA). Patients must not have unstable angina (anginal symptoms at rest) or new onset angina (began within the last 3 months) or myocardial infarction within the past 6 months.
* Prior use of sorafenib
* Known brain metastasis. Patients with neurological symptoms must undergo a CT scan/MRI of the brain to exclude brain metastasis.
* Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* Uncontrolled hypertension defined as systolic blood pressure > 150 mmHg or diastolic pressure > 90 mmHg, despite optimal medical management.
* Known human immunodeficiency virus (HIV) infection.
* Active clinically serious infection > CTCAE Grade 2 except for Except Hepatitis B(HBV) or Hepatitis C (HCV)
* Thrombolic or embolic events such as a cerebrovascular accident including transient ischemic attacks within the past 6 months.
* Serious non-healing wound, ulcer, or bone fracture.
* Evidence or history of bleeding diathesis
* Major surgery, open biopsy or significant traumatic injury within 4 weeks of first study drug.
* Use of St. John's Wort or rifampin (rifampicin).
* Known or suspected allergy to sorafenib or any agent given in the course of this trial.
* Any condition that impairs patient's ability to swallow whole pills.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09; Primary Completion 2011-05 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Adverse events associated with technical aspects of the operation | post-transplant
  To assess the safety and feasibility of treating HCC patients with sorafenib prior to OLT, as determined by the number of patients experiencing grade 4 hemorrhaging needing blood trnasfusion, thrombosis of vascular graft structures, stenosis of vascular anastomosis or biliary leaks or anastomotic biliary stenosis.

SECONDARY OUTCOMES:
Time to progression prior to OLT | 10 - 12 months
  A measure of time after being put on transplant list until the disease is beyond Milan's criteria prior to OLT.
Drop Out Rate | 10-12 months
  This is the rate of subjects who were eligible for liver transplant but drop out secondary to disease progression while awaiting donor organ.
Waiting Time | 10-12 months
  This is number of months from the time patient get listed on the transplant list to the time patient under goes actual liver transplant.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Pelley, MD, Principal Investigator — CCF Taussig Cancer Solid Tumor Oncology
Locations (1):
- Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States